CLINICAL TRIAL: NCT04746391
Title: Assessment of a Relation Between Dialyzer Clearance and Clotting in Hemodialyzer
Brief Title: Impact of Clotting on Dialyzer Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UGent_FiberClotting_2
Record Dates: First submitted 2020-09-29; First posted 2021-02-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis; Coagulation
Keywords: Hemodialyzer; Fibre Clotting
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Solacea_60min (Experimental): * blood sampling from dialyzer inlet and outlet line at 60min, just before dialysis termination
  * microCT scanning of rinsed and dried hemodialyzer, post dialysis in order to count open fibers
  Interventions: Device: Dialyzer type; Other: Dialysis duration
- Solacea_120min (Experimental): * blood sampling from dialyzer inlet and outlet line at 120min, just before dialysis termination
  * microCT scanning of rinsed and dried hemodialyzer, post dialysis in order to count open fibers
  Interventions: Device: Dialyzer type; Other: Dialysis duration
- Solacea_240min (Experimental): * blood sampling from dialyzer inlet and outlet line at 240min, just before dialysis termination
  * microCT scanning of rinsed and dried hemodialyzer, post dialysis in order to count open fibers
  Interventions: Device: Dialyzer type; Other: Dialysis duration
- FX800_60min (Experimental): * blood sampling from dialyzer inlet and outlet line at 60min, just before dialysis termination
  * microCT scanning of rinsed and dried hemodialyzer, post dialysis in order to count open fibers
  Interventions: Device: Dialyzer type; Other: Dialysis duration
- FX800_120min (Experimental): * blood sampling from dialyzer inlet and outlet line at 120min, just before dialysis termination
  * microCT scanning of rinsed and dried hemodialyzer, post dialysis in order to count open fibers
  Interventions: Device: Dialyzer type; Other: Dialysis duration
- FX800_240min (Experimental): * blood sampling from dialyzer inlet and outlet line at 240min, just before dialysis termination
  * microCT scanning of rinsed and dried hemodialyzer, post dialysis in order to count open fibers
  Interventions: Device: Dialyzer type; Other: Dialysis duration

INTERVENTIONS:
Device: Dialyzer type — Fiber blocking and dialyzer clearance is calculated in two different commercially available dialyzers
Other: Dialysis duration — Fiber blocking and dialyzer clearance is calculated for three different dialysis durations

SUMMARY:
Coagulation within the dialyzer membrane fibres is an obvious biological sign of bio-incompatibility. To avoid clotting during extracorporeal treatment, an anticoagulant is added to the circuit, resulting in an increased risk for bleeding complications. In addition, there is evidence that a substantial number of fibers can become blocked before this is reflected in routinely observed parameters, or in termination of the dialysis session. Little is known about the impact of such subclinical clotting on dialyzer performance in terms of solute clearance. Membrane clogging may influence both the diffusive and convective transport characteristics of the dialyzer membrane before leading to complete dialyzer clotting. In 2018, we described a method to objectively count the number of blocked fibres inside a dialyzer using a micro-CT scanning technique. In the present trial, we use this method to assess the number of open fibers post dialysis, and this for three different dialysis durations and in two different dialyzer types. Just before the termination of the dialysis session, dialyzer clearance is assessed for different solutes from concentration measurements in blood samples as taken from the dialyzer inlet and outlet line.

The aim of this randomized cross-over study is to objectively quantify the impact of blocked fibers on the performance of different dialyzer membranes: ATA™ (asymmetric triacetate) membrane in the Solacea™ dialyzer, and polysulfone membrane in the FX800Cordiax dialyzer, and this with a decreased anticoagulation dose.

DETAILED DESCRIPTION:
This single centre, randomized cross-over study includes ten consecutive stable chronic hemodialysis (HD) patients who experienced stable dialysis sessions during the last 4 weeks, and had no known coagulation disorder, active inflammation or malignancy. Double-needle vascular access is achieved through a native arterio-venous fistula or a well-functioning double lumen tunnelled central venous catheter. Patients are followed during 6 consecutive midweek dialysis sessions. At midweek, patients receive only 1/4th of their regular brand of Low-Molecular Weight Heparin anticoagulation at the beginning of the dialysis session. All test sessions are performed with blood flow at 300mL/min and dialysate flow at 500mL/min in post dilution hemodiafiltration (HDF) mode (substitution flow 75mL/min). Ultrafiltration rates are set according to the patient's interdialytic weight gain and clinical status.

Patients are randomized for hemodialyzer type and dialysis duration:

1. ATA™ Solacea 19H - 60min dialysis
2. ATA™ Solacea 19H - 120min dialysis
3. ATA™ Solacea 19H - 240min dialysis
4. polysulfone FX800Cordiax - 60min dialysis
5. polysulfone FX800Cordiax - 120min dialysis
6. polysulfone FX800Cordiax - 240min dialysis

Just before the termination of the 6 experimental midweek sessions, blood is sampled from the inlet and outlet blood lines. Blood samples are immediately centrifuged and serum vials are stored at -80°C until batch analysis. Post dialysis, dialyzers are rinsed and dried and scanned with micro computed tomography (CT) to count the number of open fibers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* experienced stable dialysis sessions during the last 4 weeks
* double needle/lumen well-functioning vascular access

Exclusion Criteria:

* known coagulation disorder
* active inflammation
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Fibre blocking in hemodialyzers | 6 weeks
  Fibre blocking as assessed post dialysis by a reference microCT scanning technique
Hemodialyzer performance | 6 weeks
  Dialyzer performance based on calculated clearances for different solutes

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital - Nephrology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanommeslaeghe F, Van Biesen W, Dierick M, Boone M, Dhondt A, Eloot S. Micro-computed tomography for the quantification of blocked fibers in hemodialyzers. Sci Rep. 2018 Feb 8;8(1):2677. doi: 10.1038/s41598-018-20898-w. PMID 29422614